CLINICAL TRIAL: NCT01724996
Title: Usefulness of Chest Wall Tenderness as Bedside Test to Exclude Acute Coronary Syndrome in Different Demographic Groups
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: CP1
Record Dates: First submitted 2012-11-05; First posted 2012-11-12 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Clinical examination: chest wall tenderness — The physical examination includes the testing of chest wall tenderness: Palpation of chest wall tenderness in lying 30° elevation of chest position. Flat index with standardized pressure where spontaneous maximum pain is reported (reproducible vs. not reproducible pain vs. no pain). Negative control (right side of chest mid-clavicle intercostal 6/7), reproducible vs. not reproducible pain vs. no pain.

SUMMARY:
To determine the significance of a simple bedside clinical test (chest wall tenderness) to exclude myocardial ischemia in different demographic groups.

DETAILED DESCRIPTION:
When a patient is presenting with acute chest pain at the ER of the University Hospital of Zurich, the study physician in charge, who is acting simultaneously as one of four attending clinical physicians, is performing the physical examination according to routine clinical practice. The physical examination includes the testing of chest wall tenderness: Palpation of chest wall tenderness in lying 30° elevation of chest position. Flat index with standardized pressure where spontaneous maximum pain is reported (reproducible vs. not reproducible pain vs. no pain). Negative control (right side of chest mid-clavicle intercostal 6/7), reproducible vs. not reproducible pain vs. no pain. The same physician, who is blinded for the final diagnosis at the time of the physical examination, is also recording the patient history including the study interview using the standardized study questionnaire.

ELIGIBILITY:
Inclusion criteria: All patients over the age of 18 years presenting with the leading symptom of first time or recurrent acute chest pain in the emergency room of the Department of Internal Medicine, University Hospital of Zurich.

Exclusion criteria:

* Missing informed consent.
* Cardiopulmonary unstable patients.
* No self reported chest pain.
* Recent thoracic surgery within1 year, inflammatory joint disease, fibromyalgia, cardiogenic shock.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patiens seaking the Emergency room of the University Hospital Zurich because of chest pain
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Chest wall tenderness | From first presententation to omission (6-12 hours)
  Chest wall tenderness in patients presenting with acute chest pain and acute coronary syndrome (ACS) (ST-elevation myocardial infarction, STEMI/Non-ST-elevation myocardial infarction, NSTEMI /unstable angina pectoris) vs. chest wall tenderness in patients presenting with chest pain and without ACS in different demographic groups (Age under vs. over 50 years; male vs. female, with vs. without CVRF).

SECONDARY OUTCOMES:
Pain description | 6-12 hours
  Localization/Radiation of pain/first time/recurrent/ Patient thinks heart is the cause/ different CVRF/Illicit drugs/Medication - in combination with "reproducible/not reproducible pain" associated with ACS

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Franzen, MD, Principal Investigator — University Hospital Zurich, Division of Internal Medicine
Locations (1):
- University Hospital Zurich, Division of Internal Medicine, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Grani C, Senn O, Bischof M, Cippa PE, Hauffe T, Zimmerli L, Battegay E, Franzen D. Diagnostic performance of reproducible chest wall tenderness to rule out acute coronary syndrome in acute chest pain: a prospective diagnostic study. BMJ Open. 2015 Jan 28;5(1):e007442. doi: 10.1136/bmjopen-2014-007442. PMID 25631316